CLINICAL TRIAL: NCT01415531
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of Nebivolol in Younger Patients (18 - 54 Years) Who Have Stage 1 or 2 Essential Hypertension
Brief Title: Study of the Efficacy and Safety of Nebivolol in Younger Patients (18 - 54 Years)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEB-MD-28
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-03

CONDITIONS: Hypertension
Keywords: Stage 1; Stage 2; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nebivolol (non-trade 5, 10 or 20 mg tablet), oral administration
  Interventions: Drug: Nebivolol
- 2 (Placebo Comparator): Dose-matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nebivolol — Nebivolol (non-trade 5, 10 or 20 mg tablet), oral administration
  Arms: 1
Drug: Placebo — Dose-match placebo
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and tolerability of 8 weeks of therapy with nebivolol in comparison to placebo in younger patients 18 - 54 years of age with stage 1 or stage 2 essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, of age 18 - 54 years
* Patients diagnosed with stage 1 or stage 2 essential hypertension
* Normal physical examination findings and electrocardiogram (ECG) results or abnormal findings judged by the Investigator to be not clinically significant

Exclusion Criteria:

* Secondary hypertension or severe hypertension
* History of Type 1 diabetes mellitus
* A medical contraindication to discontinuing a current antihypertensive therapy
* Clinically significant respiratory disease that prohibit use of a beta blocker

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 641 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Lukic, MD, M. Sc., Study Director — Forest Laboratories
Locations (75):
- United States (75):
  - Forest Investigative Site 065, Phoenix, Arizona
  - Forest Investigative Site 067, Phoenix, Arizona
  - Forest Investigative Site 070, Phoenix, Arizona
  - Forest Investigative Site 049, Buena Park, California
  - Forest Investigative Site 034, Burbank, California
  - Forest Investigative Site 039, Costa Mesa, California
  - Forest Investigative Site 024, Fountain Valley, California
  - Forest Investigative Site 020, Fresno, California
  - Forest Investigative Site 021, Fresno, California
  - Forest Investigative Site 040, Greenbrae, California
  - Forest Investigative Site 047, La Mesa, California
  - Forest Investigative Site 073, Los Angeles, California
  - Forest Investigative Site 077, Roseville, California
  - Forest Investigative Site 060, San Bernardino, California
  - Forest Investigative Site 054, San Francisco, California
  - Forest Investigative Site 018, Spring Valley, California
  - Forest Investigative Site 028, Denver, Colorado
  - Forest Investigative Site 059, Brooksville, Florida
  - Forest Investigative Site 033, Fort Lauderdale, Florida
  - Forest Investigative Site 006, Hallandale, Florida
  - Forest Investigative Site 044, Longwood, Florida
  - Forest Investigative Site 001, Miami, Florida
  - Forest Investigative Site 012, Miami, Florida
  - Forest Investigative Site 032, Miami, Florida
  - Forest Investigative Site 055, Miami, Florida
  - Forest Investigative Site 045, Oviedo, Florida
  - Forest Investigative Site 031, St. Petersburg, Florida
  - Forest Investigative Site 009, Atlanta, Georgia
  - Forest Investigative Site 007, Chicago, Illinois
  - Forest Investigative Site 004, Morton, Illinois
  - Forest Investigative Site 072, Evansville, Indiana
  - Forest Investigative Site 069, Newburgh, Indiana
  - Forest Investigative Site 025, Augusta, Kansas
  - Forest Investigative Site 029, Louisville, Kentucky
  - Forest Investigative Site 068, Madisonville, Kentucky
  - Forest Investigative Site 061, Metairie, Louisiana
  - Forest Investigative Site 057, New Orleans, Louisiana
  - Forest Investigative Site 058, New Orleans, Louisiana
  - Forest Investigative Site 008, Lutherville, Maryland
  - Forest Investigative Site 062, Fall River, Massachusetts
  - Forest Investigative Site 075, Paw Paw, Michigan
  - Forest Investigative Site 019, Brooklyn Center, Minnesota
  - Forest Investigative Site 017, Chaska, Minnesota
  - Forest Investigative Site 038, Belzoni, Mississippi
  - Forest Investigative Site 035, Olive Branch, Mississippi
  - Forest Investigative Site 023, Las Vegas, Nevada
  - Forest Investigative Site 048, Las Vegas, Nevada
  - Forest Investigative Site 052, Las Vegas, Nevada
  - Forest Investigative Site 014, Elizabeth, New Jersey
  - Forest Investigative Site 051, Trenton, New Jersey
  - Forest Investigative Site 003, Asheboro, North Carolina
  - Forest Investigative Site 010, Charlotte, North Carolina
  - Forest Investigative Site 011, Raleigh, North Carolina
  - Forest Investigative Site 016, Raleigh, North Carolina
  - Forest Investigative Site 005, Wilmington, North Carolina
  - Forest Investigative Site 036, Winston-Salem, North Carolina
  - Forest Investigative Site 002, Columbus, Ohio
  - Forest Investigative Site 050, Norman, Oklahoma
  - Forest Investigative Site 030, Portland, Oregon
  - Forest Investigative Site 056, Downingtown, Pennsylvania
  - Forest Investigative Site 022, Pelzer, South Carolina
  - Forest Investigative Site 053, Beaumont, Texas
  - Forest Investigative Site 066, Boerne, Texas
  - Forest Investigative Site 076, Corpus Christi, Texas
  - Forest Investigative Site 037, Dallas, Texas
  - Forest Investigative Site 043, Haltom City, Texas
  - Forest Investigative Site 015, Houston, Texas
  - Forest Investigative Site 026, Houston, Texas
  - Forest Investigative Site 027, Houston, Texas
  - Forest Investigative Site 074, Houston, Texas
  - Forest Investigative Site 071, Orem, Utah
  - Forest Investigative Site 042, Sandy City, Utah
  - Forest Investigative Site 063, Norfolk, Virginia
  - Forest Investigative Site 064, Norfolk, Virginia
  - Forest Investigative Site 046, Port Orchard, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over a 4 month period from August 2011 to December 2011 at 76 study sites in the United States.
Groups:
- Placebo: Dose-matched placebo
Period: Overall Study
Arm/Group | Placebo | Nebivolol
Started | 214 | 427
Completed | 189 | 390
Not Completed | 25 | 37
Not completed — Adverse Event | 7 | 10
Not completed — Lack of Efficacy | 3 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 6 | 14
Not completed — Lack of Compliance | 1 | 4
Not completed — Other Reasons | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nebivolol | Total
Number analyzed (Participants) | 214 | 427 | 641
Age Continuous [Mean (Standard Deviation); unit: years]
  18 to 54 | 46.0 (6.9) | 44.9 (6.9) | 45.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 190 | 285
  Male | 119 | 237 | 356
Region of Enrollment [Number; unit: participants]
  United States | 214 | 427 | 641

OUTCOME MEASURES:

1. Primary Outcome: Trough Seated Diastolic Blood Pressure (DBP)
Description: Change from baseline in mean seated trough cuff Diastolic Blood Pressure (DBP) at Week 8 as measured by an Omron device. The primary efficacy analysis was based on the Intent to Treat (ITT) population using a Last Observation Carried Forward (LOCF) approach.
Time Frame: Change from Baseline to Week 8
Population: 641 patients were randomized to receive double-blind treatment. The Safety population consisted of 641 patients who received at least 1 dose of double-blind treatment. The Intent to Treat population (ITT) consisted of 634 patients who had at least 1 postbaseline seated diastolic blood pressure (DBP) assessment
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Placebo | Nebivolol
Number analyzed (Participants) | 211 | 423
mmHG | -5.5 (9.5) | -11.8 (8.8)
Statistical Analysis 1: Comparison: Placebo vs Nebivolol; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -6.3, 95% CI 2-sided [-7.7 to -4.8]

2. Secondary Outcome: Trough Seated Systolic Blood Pressure (SBP)
Description: Change from baseline in mean seated trough cuff Systolic Blood Pressure (SBP) at Week 8 as measured by an Omron device. The secondary efficacy analysis was based on the Intent to Treat (ITT) population using a Last Observation Carried Forward (LOCF) approach.
Time Frame: Change from Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nebivolol
Number analyzed (Participants) | 211 | 423
mm Hg | -5.5 (13.9) | -13.7 (14.5)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 9 month period from August of 2011 to April of 2012
Description: The Safety population consisted of 641 randomized patients who received at least 1 dose of double-blind treatment.
Arm/Group | Placebo | Nebivolol
Serious Adverse Events (participants affected / at risk) | 4/214 | 4/427
Other Adverse Events (participants affected / at risk) | 21/214 | 37/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=214) | Nebivolol (N=427)
Hypersensitivity (Immune system disorders) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=214) | Nebivolol (N=427)
Upper respiratory tract infection (Infections and infestations) | 4 | 23
Headache (Nervous system disorders) | 17 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc